CLINICAL TRIAL: NCT00312130
Title: A Single-blind, Single-treatment Study to Evaluate the Effects of Vildagliptin on Response to an Intravenous Glucose Load in Pre-diabetic Subjects With Impaired Fasting Glucose
Brief Title: A Study to Evaluate the Effects of Vildagliptin on the Insulin Response to Glucose in Subjects With Pre-diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CLAF237A2345
Record Dates: First submitted 2006-04-06; First posted 2006-04-07 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Pre-diabetes
Keywords: Vildaglptin; Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This is an exploratory study to assess whether vildagliptin, an unapproved drug, can increase insulin secretion in subjects with pre-diabetes who have a defect in the insulin response and elevated levels of fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

* BMI in the range 22-45 and with a stable weight for the last 6 months
* Blood glucose criteria must be met
* Written informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Previous diagnosis of type 2 diabetes or treatment with hypoglycemic agents
* Type 1 diabetes
* Evidence of cardiovascular complications as defined by the protocol
* Evidence of diabetic complications as defined by the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in acute insulin response to an iv glucose load at 6 weeks

SECONDARY OUTCOMES:
Change from baseline in glucose disappearance rate at 6 weeks
Change from baseline in glucose disappearance rate at 8 weeks
Change from baseline in insulin sensitivity at 6 weeks
Change from baseline in insulin sensitivity at 8 weeks
Change from baseline in acute insulin response to an iv glucose load at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Utzschneider KM, Tong J, Montgomery B, Udayasankar J, Gerchman F, Marcovina SM, Watson CE, Ligueros-Saylan MA, Foley JE, Holst JJ, Deacon CF, Kahn SE. The dipeptidyl peptidase-4 inhibitor vildagliptin improves beta-cell function and insulin sensitivity in subjects with impaired fasting glucose. Diabetes Care. 2008 Jan;31(1):108-13. doi: 10.2337/dc07-1441. Epub 2007 Oct 1. PMID 17909087